CLINICAL TRIAL: NCT02262338
Title: A Phase 1 Safety and Dose-Finding Study of a Human Insulin Receptor Monoclonal Antibody-Human Iduronate 2-Sulfatase (IDS) Fusion Protein, AGT-182 in Adult Patients With Mucopolysaccharidosis II (MPS II, Hunter Syndrome)
Brief Title: Safety and Dose Ranging Study of Insulin Receptor MoAb-IDS Fusion Protein in Patients With Hunter Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArmaGen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGT-182-101
Record Dates: First submitted 2014-10-02; First posted 2014-10-13 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Mucopolysaccharidosis II
Keywords: MPS II; Hunter Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated subjects (Experimental): AGT-182 solution for infusion will be administered intravenously at doses of 1.0 mg/kg or 3.0 mg/kg weekly for 8-13 weeks.
  Interventions: Drug: AGT-182

INTERVENTIONS:
Drug: AGT-182 — Recombinant HIRMAb-IDS

SUMMARY:
AGT-182 is a fusion protein containing idursulfase that is intended to deliver the enzyme peripherally and to the brain, when administered intravenously. This study is a safety and dose ranging study to obtain safety and exposure data, as well as information on the biological activity of the investigational drug.

DETAILED DESCRIPTION:
This is a sequential, open-label, dose escalation, multi-dose study in adults with Hunter syndrome. Two dose levels, assuming tolerability, are planned sequentially, with safety data from the previous cohort being reviewed prior to escalation to the next higher dose cohort. Subjects will receive weekly doses of AGT-182 for 8 weeks if ERT-naive or agreeing to a 6-week ERT washout, or for 13 weeks if currently taking ERT and not agreeing to washout.

ELIGIBILITY:
Inclusion Criteria:

* Male age 18 years or older
* Diagnosis of Hunter Syndrome (documented fibroblast or leukocyte IDS enzyme activity level of less than 10% of the lower limit of the normal range of the measuring laboratory - or any level of enzyme deficiency together with the presence of a pathogenic mutation in the IDS gene - and documentation of normal enzymatic activity of at least 1 other sulfatase.)
* Must fall into one of the following groups:

  * currently receiving standard enzyme replacement therapy (ERT) and be willing to discontinue it for the study duration, taking AGT-182 instead
  * have not received standard ERT for at least 3 months and have elevated uGAGs of at least 3.5 fold above age-related normals at study screening
  * have never received ERT
* Voluntary written consent
* Sexually mature males must be advised to use a medically accepted method of contraception throughout the study.

Exclusion Criteria:

* Refusal to complete screening/baseline evaluations
* Receipt of an investigational drug within the prior 90 days
* Any medical condition or other circumstances that may significantly interfere with study compliance
* Clinically significant spinal cord compression, evidence of cervical instability
* Known hypersensitivity to idursulfase or any of the components of AGT-182
* Known to be nonresponsive to standard ERT treatment (i.e., high uGAG values despite taking full dose standard ERT)
* History of diabetes mellitus or hypoglycemia
* Contraindication to lumbar puncture, if the patient agrees to this optional assessment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
number of participants with adverse events as a measure of safety and tolerability | 8 weeks (ERT-naive) or 13 weeks (ERT)

SECONDARY OUTCOMES:
plasma pharmacokinetic parameters (maximal concentration, half-life, area under the curve, mean residence time, volume of distribution and clearance of AGT-182) | 8 weeks (ERT-naive) or 13 weeks (ERT)
change in urinary or plasma glycosaminoglycans (GAGs) | 8 weeks (ERT-naive) or 13 weeks (ERT)
change in liver or spleen size | 8 weeks (ERT-naive) or 13 weeks (ERT)
change in cerebrospinal fluid (CSF) glycosaminoglycans (GAGs) | 8 weeks (ERT-naive) or 13 weeks (ERT)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Rioux, MD PhD, Study Director — ArmaGen, Inc
Locations (5):
- United States (3):
  - Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Emory University, Decatur, Georgia
- ZKJM MC University of Mainz, Mainz, Germany
- Institute of Human Genetics, National Inst of Health, University of the Philippines, Manila, Philippines